CLINICAL TRIAL: NCT04639752
Title: Effectiveness of Remote Peer Support in Prevention of Postpartum Depression: a Randomized Controlled Trial
Brief Title: Remote Peer Support in Prevention of Postpartum Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Antonin Sebela, Principal Investigator, National Institute of Mental Health, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NU21J-09-00064
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Two groups: One receives MSM prevention intervention and the other group receives Enhanced Treatment as Usual (referral and monitoring).
Who Masked: Outcomes Assessor
Masking Description: The person administering the outcome measures is blind to participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mom´s Supporting Mom (MSM) (Experimental): A preventive intervention that involves psychoeducation and peer techniques described in study detailed description.
  Interventions: Behavioral: Mom´s Supporting Mom
- Enhanced Treatment as Usual (Active Comparator): Referral to treatment in the community and monitoring
  Interventions: Behavioral: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Mom´s Supporting Mom — A preventive peer consultation intervention for Postpartum Depression.
  Other Names: MSM
  Arms: Mom´s Supporting Mom (MSM)
Behavioral: Enhanced Treatment As Usual — Referral to treatment in the community, clinical monitoring
  Other Names: ETAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
The project aims to test the clinical effectiveness of the Mom´s Supporting Moms intervention, a newly developed approach to the prevention of postpartum depression (PPD) and to determine its cost-effectiveness. The approach consists of online screening for risk of PPD in obstetric settings, and subsequent remote peer support intervention for women at risk of PPD development. As a preparation for proposed study, investigators have developed the Mom´s Supporting Moms intervention which is based in mother-to-mother delivered psychoeducation, basic procedures of cognitive behavioral therapy and mindfulness, shared personal experience with postpartum depression and, if necessary, referring to a professional consultation. Proposed study will allow investigators to bring missing Czech methodological procedures for the early screening of PPD development risk, and for subsequent non-pharmacological intervention. Further, investigators will be able to present economic data on proposed intervention to relevant stakeholders in mental health policy.

To achieve these aims, investigators will 1) set up a screening program in five Czech maternity hospitals 2) conduct a randomized controlled trial (n= 60 per each arm), and 3) conduct a cost-effectiveness analysis of the Mom´s Supporting Moms intervention.

Investigators will test the following primary hypotheses: H1: Mom´s Supporting Moms intervention will decrease depressive symptoms in women at risk of PPD development. Secondary hypotheses: SH1: Mom´s Supporting Moms intervention will reduce anxiety symptoms in women at risk of PPD development. SH2: Mom´s Supporting Moms intervention will increase women's health-related quality of life. SH3: Mom´s Supporting Moms intervention is cost-effective in comparison to treatment as usual.

DETAILED DESCRIPTION:
RELEVANCE

Although PPD is a widespread problem that complicates not only women´s life, but also the development of the infant, which has long-term consequences on their future health and well-being, the vast majority of affected women are left untreated. PPD has been increasingly recognized as a major public health issue and there is a growing sense of urgency to identify approaches to better manage it.

In the Czech Republic, however, women themselves, their children and society do not benefit from decades of basic research on complex negative effects of postpartum mood disorders as the knowledge obtained from it has not been translated into a systematic intervention. The care of women facing postpartum mental disorders is fragmented in the Czech Republic and is not addressed systematically by a step-by-step approach. Further, there is no system in the Czech Republic for the prevention of perinatal mental disorders in women, which also plays a preventive role in the development of mental disorders in the children of these mothers.

METHODS

1. Screening Phase - identification of women at risk of PPD development Participants: Consenting women who will give a birth in maternity hospitals (Mělník, Neratovice, Bulovka, Thomayer, and Olomouc).

   Intervention: An online psychosocial risk screening software, which investigators pilot tested, will be actively offered in cooperating maternity hospitals. Consenting women will complete the online screening form, running on the servers of the National Institute of Mental Health, secured against cybercrime, before participants will leave the maternity hospital (day 3-4 after delivery).

   The screening instrument consists of the Edinburgh Postpartum Depression Scale - EPDS, Perinatal Anxiety Screening Scale - PASS, and the Perinatal Psychosocial Profile - PPP.

   The main domain of interest is the presence of depressive symptoms (EPDS), the secondary domains are the presence of anxiety symptoms (PASS) and the presence of psychosocial stress (PPP).

   After completing the screening form, participants with an EPDS score <10 will be sent an automatic email thanking participants for participating in the study and informing them of a low risk of developing PPD.

   If a participant scores ≥ 10 in the EPDS, participant will be considered as at risk of PPD development (Knights et al., 2016), and an automatic email inviting these women in the Intervention phase will be sent to these participants based on automated randomization (allocation 1:1, experimental:control):
   1. for the experimental group with the information that, based on the screening results, participants have higher risk of mental discomfort, and that participants will be contacted by a peer consultant within 2-3 days.
   2. for the control group with the information that participants have a higher risk of mental discomfort according to the screening, and therefore investigators attach information on how to proceed if participants want to actively seek care.

   The screening result of each woman with EPDS ≥ 10 who will be randomized to the intervention group will be also sent to the peer support coordinators so that the coordinator can connect the woman with the peer consultant.

   Specific situation in screening: Question EPDS 10: I had thoughts of hurting myself. If a participant answer - Yes, very often.

   Participants screening will be evaluated as high-risk and participant will be automatically connected with a peer coordinator who will offer her a professional psychiatric / psychological consultation. If that situation occurs, it will be properly recorded, and participant will be excluded from the study.
2. Intervention Phase

   - a randomized controlled trial. Participants: women at risk of PPD identified through the Screening Phase of the proposed study. Criteria for inclusion in the Intervention Phase: EPDS score ≥ 10.

   Intervention: Mom´s Supporting Moms - remote peer support. At least 4 times telephone contact (or contact via another telecommunication channel, according to the study participant's preference - Skype, Zoom, WhatsApp, Facebook Messenger, etc.) between the research participant and a peer consultant trained by the National Institute of Mental Health - Czech Republic. Within peer support, the main method is listening, psychoeducation, basic procedures of cognitive behavioral therapy and mindfulness, shared personal experience with PPD and postpartum anxiety disorders and, if necessary, referring to a professional consultation.

   Comparison: usual postpartum care consisting of gynecology check-ups which are in the Czech Republic predominantly focused on somatic health. Women have to actively seek for help if they need mental health care. Participants from the control group, who will seek themselves the Mom´s Supporting Moms intervention will be excluded from the study.

   Randomization: automatized randomization of all participants identified in the Screening Phase as being at risk of PPD development to experimental arm (Mom´s Supporting Moms intervention) or to control arm (usual postpartum care), allocation 1:1.
3. Cost-effectiveness analysis (CEA) - economy analysis of the Mom´s Supporting Moms The CEA result provides information on the cost per unit of health benefit. Economic evaluation is strictly comparative, and its purpose is always to compare the results of at least two alternative treatment approaches.

   For this reason, CEA's outputs are always relative and measure the change in costs (incremental costs) and change in benefits (incremental effects) given by using one alternative instead of another. The incremental cost-effectiveness ratio (ICER) is defined as the change in the average costs of an alternative divided by the change in average benefits, and very often investigators compare a new treatment with an existing treatment:

   The costs of the monitored treatment strategies are obtained by weighing the services provided to the patient for the year of monitoring by their price, i.e. by multiplying the quantity of the provided service by the unit value of the given service. The Czech Republic has rich national registers of administrative data on the use of health services. In 2016, the National Register of Paid Health Services (NRHZS) was newly established, which collects data on the use of inpatient and outpatient services and on the consumption of medicines by all insured persons. Investigators will calculate the final prices on the basis of the payment decree. The value of the peer intervention will be quantified and included in the ICER calculation.

   Linking a clinical dataset to registry data: To perform the CEA, investigators will link clinical data from the intervention part of the study with data from the NRHZS, which has been managed by the Institute of Health Information and Statistics of the Czech Republic since 2016.
4. Analytic plan Primary outcome is the between group (experimental arm vs. control arm) difference in Edinburgh Postnatal Depression Scale in week 6. Investigators will use ANCOVA test (difference in post- intervention score wit baseline score as covariate) to test the effect of intervention on the self-reported depressive symptoms. Intention-to-treat analysis will be used with the last value observed carried forward method used for missing observations. Investigators will adjust for confounders (possibly: age, marital status, childbirth complications, psychosocial stress) if between group differences in these variables will be observed. For the secondary outcomes (Perinatal Anxiety Screening Scale - anxiety symptoms and AQoL-8D - quality of life) investigators will use similar statistical approach as described in the analytic plan for the primary outcome.

   The between group differences in the distribution of mental disorders assessed by the MINI interview postintervention (week 6, month 3 after randomization) will be tested by the chi-square tests and presented as the RRs with 95% CI. Exploratory analysis: Investigators will use a repeated measures analysis using a linear mixed model to assess the trend of the examined outcomes over the period of 3 months. The interaction effect of group and time will be used to assess the differences over time.

   The CEA: The effectiveness Mom´s Supporting Moms will be measured by the quality-adjusted life-years (QALYs) determined by the AQoL-8D data measured baseline, week 6, month 3 and year 1 after randomization. Investigators will use the standard area under the curve method to calculate QALYs. The estimation of costs of health-care services and medication use will be done according to appropriate Czech payment decree. Further, investigators will divide differences in costs during the follow-up period between the two groups by differences in QALYs to estimate the incremental costeffectiveness ratio (ICER). Then the cost-effectiveness plane will be produced (i.e., a diagram with difference in QALYs on the horizontal axis and difference in costs on the vertical axis displaying the central cost-effectiveness estimate and the uncertainty in terms of these two dimensions). Finally, investigators will calculate the cost-effectiveness acceptability curve that, in our case, will shows the estimated probability that intervene by Mom´s supporting Moms is cost-effective given the sampling uncertainty. A regression approach will be used for our analyses if any confounders will be detected.
5. Power analysis - estimated for our primary outcome According to previously published studies, the effect of peer support in reducing the rate of self-assessed depressive symptoms is moderate. The sample size is calculated so that investigators can detect a medium-sized intergroup difference on the Edinburgh Postnatal Depression Scale (effect size 0.6) at a power of 80% and a significance level of 5% (2-sided). Thus, with the power analysis set in this way and a potential drop out of 30%, the minimum file size included in the intervention part of the study is 120 women (60 for each group).

ELIGIBILITY:
SCREENING PHASE

Criteria for inclusion:

* sex-female
* childbirth in the hospital
* signing of informed consent
* email address ownership
* age 18 - 45 years

Exclusion Criteria:

- acute medical illness or significant pregnancy complication (based on self-report)

INTERVENTION PHASE

Criteria for inclusion:

* Edinburgh Postpartum Depression Scale score ≥10.
* participant identified through the Screening Phase of the study

Exclusion Criteria:

- acute suicidal behavior (based on self-report)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Postpartum depressive symptoms | 6 weeks postpartum
  self-rated depressive symptomatology measured by Edinburgh Postnatal Depression Scale. Score range 0-30, higher score represents worse outcome.

SECONDARY OUTCOMES:
Postpartum anxiety symptoms | 6 weeks postpartum
  self-rated anxiety symptomatology measured by Perinatal Anxiety Screening Scale. Score range 0-93, higher score represents worse outcome.
Postpartum health-related quality of life | 6 weeks postpartum
  self-rated health-related quality of life measured by Assessment of Quality of Life- 8 dimensions. Score range 0 - 177, higher score represents worse outcome.
Cost-effectiveness | 6 weeks, 3 months, and year 1 postpartum
  The effectiveness Mom´s Supporting Moms will be measured by the quality-adjusted life-years (QALYs) determined by the AQoL-8D data. The estimation of costs of health-care services and medication use will be done according to appropriate Czech payment decree.

OTHER OUTCOMES:
Postpartum depressive symptoms | 3 months postpartum
  self-rated depressive symptomatology measured by Edinburgh Postnatal Depression Scale. Score range 0-30, higher score represents worse outcome.
Postpartum anxiety symptoms | 3 months postpartum
  self-rated anxiety symptomatology measured by Perinatal Anxiety Screening Scale. Score range 0-93, higher score represents worse outcome.
Postpartum health-related quality of life | 3 months postpartum
  self-rated health-related quality of life measured by Assessment of Quality of Life- 8 dimensions. Score range 0 - 177, higher score represents worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Antonin Sebela, Ph.D., Principal Investigator — National Institute of Mental Health, Klecany, Czechia
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be made available to other researchers.
Supporting Information: ICF
Time Frame: After the completion of the study
Access Criteria: Permission of the PI

REFERENCES:
- [Derived] Sebela A, Horakova A, Nemcova H, Kuklova M, Noskova E, Svancer P, Byatt N, Janovska A, Hrdlickova K. Mom Supporting Mom: Effective Peer Support Intervention for Women with Postpartum Psychological Distress. Psychosoc Interv. 2025 Jul 29;34(3):151-160. doi: 10.5093/pi2025a12. eCollection 2025 Sep. PMID 40765646